CLINICAL TRIAL: NCT02410252
Title: Use Feasibility of the iThermonitor in Pediatric Patients on Myelosuppresive Therapies for Acute Leukemia and Other Childhood Cancers
Brief Title: Use Feasibility of the iThermonitor in Pediatrics Patients on Myelosuppresive Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-485
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myeloid Leukemia; Non-Hodgkin Lymphoma
Keywords: continuous temperature monitoring; patient self-management; iThermonitor; Home monitoring
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iThermonitor (Experimental): Participants are asked to use the iThermonitor device for two weeks to monitor their temperature. Participants are asked to wear the device for as many hours as they can but at a minimum to wear while sleeping.
  Interventions: Device: iThermonitor

INTERVENTIONS:
Device: iThermonitor — The device is a continuous temperature monitoring tool for home monitoring of temperature. Participants are asked to use this device for two weeks.

SUMMARY:
This is a pilot study to evaluate the use feasibility of the iThermonitor, a continuous temperature monitoring device, as a clinical support and patient self-management tool in the management of pediatrics patients on myelosuppressive therapies for acute leukemia and other childhood cancers.

DETAILED DESCRIPTION:
Neutropenia, secondary to myelosupressive therapies, predisposes patients to significant risk for infectious complications which increases morbidity and mortality. Usually, fever is the first clinical sign of the inflammatory response to the infective process; and early detection is an indication for empiric antimicrobial therapy and further evaluation to determine risk for sepsis. Today, broad-spectrum antimicrobial therapy at the first detection of fever has helped significantly decreased the mortality associated with neutropenia in the intensive phase of chemotherapy. Therefore, early detection of fever, through regular temperature monitoring, in a neutropenic patient is critical to improved clinical outcome. Vigilance on the part of care providers and care givers is crucial to early detection. Traditionally, this is simply done through episodic oral or axillary monitoring of temperature. In this study, we propose to test the use feasibility of an innovative device that continuously monitors body temperature as a clinical decision support tool in pediatric patients undergoing myelosuppressive therapies for acute leukemias and other childhood cancers.

The iThermonitor, a FDA class II device, is a high accuracy device that continuously monitors body temperature and connects to a receiver (iPad mini) via bluetooth to display body temperature data in real time. The iThermonitor is attached to the skin by a hydrogel dressing which can be changed as needed. It captures data even without connection to a receiver and it can establish connection to a paired receiver device (the iPad mini) within a range of three meters. The provided iPad mini will be pre-loaded with the iThermonitor app which will be used to pair the receiver with the iThermonitor device. The device monitors body temperature every four seconds and is able to store 10 days worth of data that can be offloaded as soon as it establishes connection with a receiver. It is able to measure temperature in the range of 25-45 degrees Celsius. Users are able to set temperature limits at which alerts for which out-of-range temperature can go off. It also provides care providers an opportunity to remotely monitor their patients' temperature in the immediate period after discharge from the hospital. Therefore, we hypothesize that the iThermonitor can serve as a feasible clinical decision support in the management of pediatric patients undergoing intensive treatments for acute leukemia and other childhood cancers.

This study will be implemented as a pilot study to test the use feasibility of the iThermonitor as a clinical decision support for continuous temperature monitoring in a dyad of 25 pediatrics patients, (aged 2yrs - 17yrs) on myelosuppressive therapies for acute leukemia and other childhood cancers at the MGH Pediatric Hematology and Oncology group, and their caregivers. The iThermonitor will be used by patients and their caregivers at home over a 2-week study period starting from the day after chemotherapy. There will be two study visits: study enrollment and study closeout.

The investigators have chosen to implement this study as a feasibility study because the investigators' goal is to determine if continuous temperature monitoring by the iThermonitor can work in home settings. To the investigators' knowledge, the researchers are not aware of any previous research exploring continuous temperature monitoring in pediatric oncology patients on myelosuppresive therapies. Therefore, findings from this study have the potential to advance knowledge about the management of fever in pediatric patients on myelosuppresive therapies.

ELIGIBILITY:
Inclusion Criteria:

* Dyad consists of a pediatric patient aged 2-17 years undergoing myelosuppressive therapies for acute leukemias and other childhood cancers.
* Dyad also includes a caregiver, ≥ 18 years of age that is willing to participate in the study.
* Ability of caregiver or patient (if old enough) to read and speak English.
* If applicable, willingness of the patient to shave axillary (armpit) hair.
* Caregiver (parent or legal guardian) must give informed consent for dyad participation.

Exclusion Criteria:

* Patient has a history of allergy to hydrogel dressing or ongoing skin diseases
* Patients with ongoing febrile illness or documented infectious disease.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Agboola, MD, MPH, Principal Investigator — Partners Connected Health Innovations
Locations (1):
- Amanda Centi, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Kakarmath SS, de Redon E, Centi AJ, Palacholla R, Kvedar J, Jethwani K, Agboola S. Assessing the Usability of an Automated Continuous Temperature Monitoring Device (iThermonitor) in Pediatric Patients: Non-Randomized Pilot Study. JMIR Pediatr Parent. 2018 Dec 21;1(2):e10804. doi: 10.2196/10804. PMID 31518304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescent-Caregiver dyads were recruited from the MGH Pediatric Cancer Center or the MGH Hospital for Children (Surgical Division). Recruitment began in early 2015 and was completed by April of 2017.
Groups:
- Temperature Monitoring Group: This was a single arm usability and feasibility study. All participants were enrolled into the same group and used the temperature monitoring device for 2 weeks.
Period: Overall Study
Arm/Group | Temperature Monitoring Group
Started | 25
Completed | 19
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- Temperature Monitoring Group: This was a single arm usability and feasibility study. All participants were enrolled into the same group where they used the study device to monitor their temperature for two weeks.
Arm/Group | Temperature Monitoring Group
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 8 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19
Age of Caregivers [Mean (Standard Deviation); unit: years] | 41 (8)
Employment Status of Caregivers [Count of Participants; unit: Participants]
  Employed, full time | 5
  Employed, part time | 3
  Homemaker | 6
  Unemployed | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants That Successfully Used the iThermonitor
Description: This will be assessed by ability of the device to successfully capture, transmit and display the patient's body temperature data on the study iPod TouchiPad mini. To limit recall bias, subjects will be required to log the ability to view the temperature data on the iPad mini once a day for the entire duration of the study. The device will be deemed a feasible continuous temperature monitoring tool if at least 80% of study subjects are able to successfully use the iThermonitor to monitor their body temperature. A subject must be able to view temperature data on the provided iPad mini at least 80% of the time in the study to be considered successful. "Time in the study" here is defined as the number of days the subject spends in the study which is expected to be two weeks.
Time Frame: Two Weeks
Population: Caregivers of participants using the device
Measure: Number; unit: % of participants
Groups:
- Temperature Monitoring Group: This was a single arm usability and feasibility study. All participants were enrolled into the same group and monitored their body temperature using the study device for 2 weeks.
Arm/Group | Temperature Monitoring Group
Number analyzed (Participants) | 19
% of participants
  View data at least once per day | 100
  Reported receiving out of range alerts | 75
  Reported receiving 3 or more out of range alerts | 63
Statistical Analysis 1: Comparison: Temperature Monitoring Group; Descriptive statistics were used to characterize the study sample, and survey responses; Test type: Other; descriptive analysis — There was no statistical analysis conducted on demographic characteristics or baseline surveys; % = 100
Statistical Analysis 2: Comparison: Temperature Monitoring Group; Only percent will be calculated. No statistical analysis will be conducted; Test type: Other — Only percents were calculated, no formal statistical analysis was completed; Statistical analysis was not completed. This was a feasibility study with small n and was not powered to determine statistical significance; No statistical analysis was conducted as part of this study

2. Secondary Outcome: Care Giver Anxiety
Description: The Generalized Anxiety Disorder, 7 item questionnaire was given to caregivers to see if using the device increased feelings of anxiety. This will be assessed using the GAD-7 questionnaire administered at enrollment and closeout
Time Frame: 0 & 2 weeks
Population: Caregivers of participants using the device.
Measure: Count of Participants; unit: Participants
Groups:
- Temperature Monitoring Group: This was a single arm usability and feasibility study. All participants were enrolled into the same group and used the study device to monitor body temperature for 2 weeks.
Arm/Group | Temperature Monitoring Group
Number analyzed (Participants) | 19
Participants
  GAD Score_0 Weeks: No anxiety | 12
  GAD Score_0 Weeks: Mild anxiety | 3
  GAD Score_0 Weeks: Moderate anxiety | 1
  GAD Score_0 Weeks: Severe anxiety | 3
  GAD Score_2 Weeks: No anxiety | 16
  GAD Score_2 Weeks: Mild anxiety | 2
  GAD Score_2 Weeks: Moderate anxiety | 0
  GAD Score_2 Weeks: Severe anxiety | 1
Statistical Analysis 1: Comparison: Temperature Monitoring Group; GAD-7 scores were coded as a categorical variable as follows: mild anxiety (total score 0 to 5) and moderate/ severe anxiety (total score 6-15). Proportion of participants with mild and moderate/ severe anxiety at enrollment and closeout was compared using Cochran's Q test; Test type: Other; p = 0.13, Cochran-Mantel-Haenszel — Significance was set at p<0.05; % = 0.29

3. Secondary Outcome: Usability, Acceptability and Satisfaction
Description: This will be assessed by questionnaires specifically designed for this study. We will be assessing ease of use, acceptability, connection and use problems like the device falling off the skin, usefulness of out-of-range temperature alerts and adverse reactions. We will also assess to see if the device helps to build caregiver self-efficacy skills in caring for the patient.
Time Frame: 2 weeks
Population: Caregivers of participants using the device.
Measure: Count of Participants; unit: Participants
Groups:
- Temperature Monitoring Group: This was a single arm usability and feasibility study. All participants were enrolled into the same group and asked to monitor their body temperature for 2 weeks using the study device.
Arm/Group | Temperature Monitoring Group
Number analyzed (Participants) | 19
Participants
  Satisfied with ease of use of device: Definitey True | 8
  Satisfied with ease of use of device: Mostly True | 9
  Satisfied with ease of use of device: A little true | 0
  Satisfied with ease of use of device: Not true | 2
  Easy to learn to use device: Definitey True | 13
  Easy to learn to use device: Mostly True | 6
  Easy to learn to use device: A little true | 0
  Easy to learn to use device: Not true | 0
  Felt comfortable using device: number analyzed (Participants) | 18
  Felt comfortable using device: Definitey True | 13
  Felt comfortable using device: Mostly True | 3
  Felt comfortable using device: A little true | 1
  Felt comfortable using device: Not true | 1
  Able to easily monitor temperature by using device: Definitey True | 12
  Able to easily monitor temperature by using device: Mostly True | 3
  Able to easily monitor temperature by using device: A little true | 2
  Able to easily monitor temperature by using device: Not true | 2
  Feel confident monitoring temperature with device: number analyzed (Participants) | 18
  Feel confident monitoring temperature with device: Definitey True | 10
  Feel confident monitoring temperature with device: Mostly True | 4
  Feel confident monitoring temperature with device: A little true | 2
  Feel confident monitoring temperature with device: Not true | 2
  Device helpful stating discussions with doctor: number analyzed (Participants) | 17
  Device helpful stating discussions with doctor: Definitey True | 5
  Device helpful stating discussions with doctor: Mostly True | 2
  Device helpful stating discussions with doctor: A little true | 5
  Device helpful stating discussions with doctor: Not true | 5
  Using device makes me feel more connected to team: Definitey True | 2
  Using device makes me feel more connected to team: Mostly True | 7
  Using device makes me feel more connected to team: A little true | 4
  Using device makes me feel more connected to team: Not true | 6
  Would recommend device: Definitey True | 10
  Would recommend device: Mostly True | 5
  Would recommend device: A little true | 2
  Would recommend device: Not true | 2
  Found app very useful in monitoring temperature: Definitey True | 10
  Found app very useful in monitoring temperature: Mostly True | 4
  Found app very useful in monitoring temperature: A little true | 4
  Found app very useful in monitoring temperature: Not true | 1
  Found out-of-range temp alert function useful: Definitey True | 5
  Found out-of-range temp alert function useful: Mostly True | 5
  Found out-of-range temp alert function useful: A little true | 5
  Found out-of-range temp alert function useful: Not true | 4
Statistical Analysis 1: Comparison: Temperature Monitoring Group; Descriptive statistics were used to characterize the study sample, and survey responses. All analysis was conducted using STATA version 14.2 with an alpha of 0.05 set a priori. Since this was an exploratory study with descriptive statistics, a complete case analysis approach was adopted for this study; Test type: Other; p = 0.05, descriptive analysis; % = 84

ADVERSE EVENTS:
Time Frame: Adverse event information was collected during active enrollment in the study and reported annually to the IRB (over 3 years).
Groups:
- Temperature Monitoring Group: Single group subjects that will use the iThermonitor device to collect temperature information for two weeks.
  iThermonitor: The device is a continuous temperature monitoring tool for home monitoring of temperature
Arm/Group | Temperature Monitoring Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
One major limitation of our study is the lack of a control group that used another temperature measurement device such as a digital thermometer without a companion app or automated temperature measurement features.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT02410252/Prot_SAP_000.pdf